CLINICAL TRIAL: NCT06335472
Title: Ultrasound-guided Effect of Three Nerves Pulsed Radiofrequency Versus Supra-scapular Nerve Pulsed Radiofrequency Both Combined With Hydro-dissection in Reducing the Intensity of Pain in Adhesive Capsulitis
Brief Title: Three Nerves Versus Suprascapular Nerve Radiofrequency Combined With Hydrodissection in Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safa Sayed Noaman, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Three nerves radiofrequency
Record Dates: First submitted 2024-03-17; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Analgesia
Keywords: shoulder pain
MeSH Terms: conditions — Agnosia; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Ultrasound-guided effect of three nerves pulsed radiofrequency versus supra-scapular nerve pulsed radiofrequency both combined with hydro-dissection in reducing the intensity of pain in adhesive capsulitis
Who Masked: Participant, Investigator
Masking Description: pain control and range of motion in adhesive capsulitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three nerves pulsed radiofrequency with hydrodissection (Active Comparator): suprascapular nerve ,axillary nerve, lateral pectoral nerve pulsed radiofrequency combined with hydrodissection in adesive capsultis
  Interventions: Procedure: 3 nerves pulsed radiofrequency with hydrodissection
- suprascapular nerve pulsed radiofrequency with hydrodissection (Active Comparator): suprascapular nerve pulsed radiofrequency combined with hydrodissection
  Interventions: Procedure: suprascapular nerve pulsed radiofrequency with hydrodissection

INTERVENTIONS:
Procedure: 3 nerves pulsed radiofrequency with hydrodissection — Patient will be in a sitting position, targeting the SSN, needle will be pushed towards floor of the suprascapular fossa, SSN is just adjacent to the suprascapular artery.
  The axillary nerve, between the deltoid muscle posteriorly, triceps muscle caudally and humerus anteriorly, axillary nerve appears as hyperechoic round in relation to posterior circumflex humeral artery.
  Lateral pectoral nerve, middle of coracoid process should be targeted, lie within hyperechoic fascial plane between pectoralis major and pectoralis minor muscle.
  hydrodissection, US transducer will be positioned inferior to scapular line , landmarks are contours of glenoid rim and humeral head, needle will be advanced until enter the GHJ capsule.
  A solution composed of 3 mL of lidocaine 1%, 3 mL of bupivacaine 0.25%, and 1 mL of dexamethasone 40 mg, followed by infusion of up to 40 mL of normal saline, until capsule is adequately distended and resistance felt
  Other Names: radiofrequency
  Arms: three nerves pulsed radiofrequency with hydrodissection
Procedure: suprascapular nerve pulsed radiofrequency with hydrodissection — The patient will be positioned in a sitting position, PRF needle will be pushed forward towards the floor of the suprascapular fossa the SSN will be visualized just adjacent to the suprascapular artery.
  hydrodissection will be done under all aseptic measures ,the US transducer will be positioned just inferior to the scapular line , landmarks are contours of posterior glenoid rim and humeral head, needle will be advanced until the needle tip will enter the GHJ capsule.
  A solution composed of 3 mL of lidocaine 1%, 3 mL of bupivacaine 0.25%, and 1 mL of dexamethasone 40 mg, followed by an infusion of up to 40 mL of normal saline , until the capsule is adequately distended and resistance will be felt.
  Arms: suprascapular nerve pulsed radiofrequency with hydrodissection

SUMMARY:
comparison between effect of three nerves pulsed radiofrequency combined with hydro-dissection versus suprascapular nerve Pulsed Radiofrequency combined with hydrodissection on pain control in adhesive capsulitis within six months follow up.

DETAILED DESCRIPTION:
comparison between effect of three nerves suprascapular,axillary,lateral pectoral nerves pulsed radiofrequency combined with hydro-dissection versus suprascapular nerve Pulsed Radiofrequency combined with hydrodissection on pain control in adhesive capsulitis within six months follow up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients aged 30-80 years old 2. Shoulder pain existing for more than one month and reduction range of motion in at least two planes (flexion, abduction, external rotation…)

Exclusion Criteria:

1. Patient refusal
2. malignancy
3. Pre-existing neurological deficits or neuropathy
4. Significant concomitant shoulder pathology as instability of shoulder joint, labral tears, labral tears, rotator cuff calcific tendinopathy, infectious arthritis, and rheumatological disease of the shoulder
5. Previous history of fracture or shoulder dislocation, or cerebrovascular accidents.
6. Known allergic history to local anesthetic
7. Known contraindications to peripheral nerve block, including local skin infections in the block procedure area, bleeding diathesis, and coagulopathy.

   -

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
The most effective modality on pain management of shoulder adhesive capsulitis using visual analog score. | 6 month
  effect of pulsed radiofequency in reducing pain in patients suffer from adesive capsulitis

CONTACTS AND LOCATIONS:
Overall Officials: ekram osman, professor, Study Director — Assiut University
Locations (1):
- Assiut university Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided

REFERENCES:
- [Background] 3. Ruiz Ibán MA, García Navlet M, Ávila Lafuente J, Alonso Güemes S. Adhesive Capsulitis. In: Textbook of Musculoskeletal Disorders. Springer; 2023. p. 615-26.
- [Background] 3. Ruiz Ibán MA, García Navlet M, Ávila Lafuente J, Alonso Güemes S. Adhesive Capsulitis. In: Textbook of Musculoskeletal Disorders. Springer; 2023. p. 615-26. 4. Schiltz M, Goudman L, Moens M, Jo N, Hatem SM. The diagnostic value of physical examination tests in adhesive capsulitis: a systematic review. Eur J Phys Rehabil Med. 2023;59(6):724 5. Silva R, Pimentel A, Gutierres M. A literature review of the treatment options for Idiopathic Adhesive Capsulitis of the Shoulder. Orthop Spo Med Op Acc J. 2021;4:460-8. 6. . Laumonerie P, Dalmas Y, Tibbo ME, Robert S, Faruch M, Chaynes P, et al. Sensory innervation of the human shoulder joint: the three bridges to break. J Shoulder Elb Surg. 2020;29(12):e499-507. 7. Martínez-Gago A, García-Mesa Y, Cuendias P, Martín-Cruces J, Abellán JF, García-Suárez O, et al. SENSORY INNERVATION OF THE HUMAN SHOULDER JOINTS IN HEALTHY AND IN CHRONIC PAIN SHOULDER SYNDROMES. Ann Anatomy-Anatomischer Anzeiger. 2023;152206. 8. Bongiorno G, Bednarova R, Biancuzzi H, Dal Mas F, Rizzardo A, Tomasi A, et al. Pulsed Radiofrequency as a Standalone Treatment for Adhesive Capsulitis. Surgeries. 2023;4(3):335-41. 9. Eckmann MS, Johal J, Bickelhaupt B, McCormick Z, Abdallah RT, Menzies R, et al. Terminal sensory articular nerve radiofrequency ablation for the treatment of chronic intractable shoulder pain: a novel technique and case series. Pain Med. 2020;21(4):868-71. 10. Pushparaj H, Hoydonckx Y, Mittal N, Peng P, Cohen SP, Cao X, et al. A systematic review and meta-analysis of radiofrequency procedures on innervation to the shoulder joint for relieving chronic pain. Eur J Pain. 2021;25(5):986-1011. 11. Küçükbingöz, Çağatay, Bahşi, A., Bayram, T., Marufoglu , F., & Özbek, H. T. (2023). Comparison of the Effectiveness of Pulse Radiofrequency in the Treatment of Suprascapular Nerve in Chronic Shoulder Pain. European Journal of Therapeutics, 29(3), 334-340. 12. Paruthikunnan SM, Shastry PN, Kadavigere R, Pandey V, Karegowda LH. Intra-articular steroid for adhesive capsulitis: does hydrodilatation give any additional benefit? A randomized control trial. Skeletal Radiol. 2020;49:795-803. 13. Chen Y-C, Shen S-H, Chiou H-J, Wan Y-L. Management of Patients with Adhesive Capsulitis via Ultrasound-Guided Hydrodilatation without Concomitant Intra-Articular Lidocaine Infusion: A Single-Center Experience. Life. 2022;12(9):1293. 14. Faul, F., Erdfelder, E., Lang, A.-G. & Buchner, A. (2007). G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods, 39, 175-191. 15- Mousa, H. (2022): Adhesive Capsulitis Motor and Sensory Stimulation during Radiofrequency Treatment. Saudi J Med. Oct, 2022; 7(10): 549-554. 16- Shafshak TS, Elnemr R. The visual analogue scale versus numerical rating scale in measuring pain severity and predicting disability in low back pain. JCR J Clin Rheumatol. 2021;27(7):282-5.
- [Result] Leafblad N, Mizels J, Tashjian R, Chalmers P. Adhesive Capsulitis. Phys Med Rehabil Clin N Am. 2023 May;34(2):453-468. doi: 10.1016/j.pmr.2022.12.009. Epub 2023 Feb 28. PMID 37003663
- [Result] Sarasua SM, Floyd S, Bridges WC, Pill SG. The epidemiology and etiology of adhesive capsulitis in the U.S. Medicare population. BMC Musculoskelet Disord. 2021 Sep 27;22(1):828. doi: 10.1186/s12891-021-04704-9. PMID 34579697